CLINICAL TRIAL: NCT06763822
Title: Evaluation of Treatment Effect in Patients with Dry Eye Combined with Asthenopia.
Brief Title: Dry Eye and Asthenopia Treatment Effect Evaluation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2024-0089
Record Dates: First submitted 2024-12-23; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-01

CONDITIONS: Dry Eye; Asthenopia
MeSH Terms: conditions — Dry Eye Syndromes; Asthenopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dry eye (Experimental)
  Interventions: Behavioral: close eyes; Behavioral: cold compress
- non-dry eye group (Placebo Comparator)
  Interventions: Behavioral: close eyes; Behavioral: cold compress

INTERVENTIONS:
Behavioral: close eyes — ask participants to close their eyes for rest
Behavioral: cold compress — cold compress on participants' eyes for rest

SUMMARY:
Asthenopia is a group of syndroms in which the human eye can see more than its visual function can bear due to various causes, resulting in visual disorders, eye discomfort or systemic symptoms after the use of the eyes, and thus can not perform visual work normally, including pain around the eyes and orbit, blurred vision, dry eyes, tears, etc. In severe cases, headache, nausea, vertigo, etc. Belonging to a group of fatigue syndromes, has become a common problem plaguing contemporary people. The International Tear Film and Ocular Surface Association (TFOS) reported in April 2023 that the incidence of digital ocular tension is as high as 97%. Refractive errors, presbyopia, eye surgery, long-term use of video terminals and dry eyes are the main causes of visual fatigue. But for a long time, the study of visual fatigue relies more on subjective questionnaires and lacks objective indicators. The ciliary muscle of the eye is an important target for improving the regulation function, and it is also a key part affecting visual fatigue. The abnormal regulation of the ciliary muscle is considered to be involved in the mechanism of visual fatigue. accommodative microfluctuations (AMFs) are the uncontrolled fluctuations of the human eye when it fixates on a stationary object or visual icon, with a range of about 0.10D to 0.50D. It is divided into low frequency component (LFC, <0.6Hz) and high frequency component (HFC, 1.0-2.3Hz). The low frequency component is considered to be the adjustment of different focusing distances. The high frequency part is the shaking of the lens, representing the tremor of the ciliary muscle. Literature studies have shown that HFC may be an objective indicator of visual fatigue, and higher HFC usually represents visual fatigue.

According to the report of TFO DEWS II (New International Consensus on Dry Eye), dry eye is defined as a multifactorial ocular surface disease, characterized by the imbalance of tear film structure and function, accompanied by tear film instability, elevated tear osmotic pressure, ocular surface inflammation and damage, abnormal neurosensory function and other symptoms. Dry eye with asthenopia is the most common mixed asthenopia, and the symptoms are more severe. Factors such as astigmatism and refractive correction affect tear film adhesion, resulting in uneven distribution of tear film and shortening of tear film. Poor tear film quality will affect the retinal image quality, the eye to correct this retinal imaging ambiguity and efforts to adjust, long-term impact will appear visual fatigue, tear film instability and visual fatigue affect each other, forming a vicious cycle. Studies have shown that dry eye patients with short tear film rupture time (BUT) are more likely to complain of visual fatigue, and their HFC and visual function are worse. With the improvement of BUT after treatment, the symptoms of dry eye and visual fatigue are reduced, and HFC and visual fluctuation are improved, which proves the possible relationship between HFC and short BUT dry eye.

We hope to conduct a study on HFC in patients with dry eye accompanied by visual fatigue symptoms, clarify the correlation between HFC and different symptoms, signs, severity, and classification of dry eye symptoms, determine whether HFC can be used as one of the indicators of diagnosis and prognosis of dry eye disease, and depict the curve of visual fatigue and working time in different populations. The aim is to provide a new idea for clinical treatment of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* have basic reading comprehension skills and to be older than 18 years old. not have myopia degree exceeding -6.0D, hyperopia exceeding +2.0D, astigmatism degree exceeding 2.0D, or anisometropia exceeding 2.0D

Exclusion Criteria:

* presbyopia or decreased regulation function, ocular inflammation and disease, worn contact lens within 1 month, history of eye surgery within 6 months, lactating or pregnant woman, have severe systemic diseases.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2024-06-16 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
HFC (high frequency component) | 1 hour
  This study enrolled a total of 27 volunteers with dry eye and 28 volunteers without dry eye. Participants were instructed to read the text content on a tablet computer at a distance of 33.3 cm for 40 min. We measured the high-frequency components (HFC) of accommodation microfluxations to indicate the degree of asthenopia before reading, 10 minutes, 20 minutes, and 40 minutes after reading, respectively to draw the excitation curve. While detecting the recovery curve, we reorganize the participants into closed eye rest group (of 29 participants) and cold compress rest group (of 26 participants). We measured the HFC after 40 minutes of reading as starting point, and then measured the HFC after 5minutes and 15minutes of rest to draw the recovery curve.We conducted linear regression analysis to detect the high-risk factors related to asthenopia.
  Two dominant frequencies were revealed by power spectrum analysis of the microfluctuations waveform, including a low-frequency component (LFC) of

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine (SAHZU), Hangzhou, Zhejiang, China